CLINICAL TRIAL: NCT00428246
Title: Anti-Inflammatory and Endothelial Protectant Effects of Paricalcitol
Brief Title: Study of Protective Effects of Paricalcitol on Inner Layer of Vessels and Its Protective Effect on Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Abbott (Industry)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 0510-04
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Kidney Disease; Endothelial Dysfunction; Inflammation; Hypertension
Keywords: Chronic Kidney Disease; Endothelial dysfunction; Inflammation; Hypertension; paricalcitol; Blood pressure; Vitamin D; Glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation; Hypertension | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 1 mcg paricalcitol
  Interventions: Drug: paricalcitol
- 2 (Active Comparator): 2 mcg paricalcitol
  Interventions: Drug: paricalcitol
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paricalcitol — 1 mcg or 2 mcg for 4 weeks.
  Other Names: Zemplar
  Arms: 1; 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The study is about possible protective effects of paricalcitol (Zemplar) upon inflammation, blood pressure and kidney function. Kidney Inflammation occurs when white blood cells become abnormally stimulated and accumulate in the kidney and cause damage to the kidney. The purpose of this study is to determine if paricalcitol helps improve kidney injury, blood pressure control and kidney function in patients with chronic kidney disease. The study will last about 7 weeks and involves about 8 visits to the medical center.

DETAILED DESCRIPTION:
We hypothesize that use of paricalcitol in patients with chronic kidney disease will lead to improvement in oxidative stress, inflammation, endothelial function and subsequently ambulatory blood pressures and glomerular filtration rate. We will pursue our hypothesis by the three specific aims:

Aim 1: To compare oxidative stress markers in patients treated with paricalcitol before and after the study. Aim 2: To measure endothelial function by flow mediated dilation in patients with chronic kidney disease before and after paricalcitol. Aim 3: To measure actigraphy guided ambulatory blood pressure and GFR in the absence of changes in anti-hypertensive medications in patients with chronic kidney disease.

The study will be double blind randomized pilot trial in 24 patients with chronic kidney disease with 1:1:1 allocation to paricalcitol 1 microgram: paricalcitol 2 microgram: Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease with estimated GFR of 30 mL/minute or more.
* Patients receiving stable dose of ACE inhibitor or Angiotensin receptor blockers for at least one month.
* Patients not currently hypertensive more than 180/110 mmHg by clinic blood pressure.
* Hemoglobulin A1C< 11%

Exclusion Criteria:

* Patients taking vitamin D analogs
* Calcium> 10 mg/dL
* Phosphorus>6 mg/dL
* Patients with anticipated need of dialysis in the next 6 weeks
* Patients unstable in the opinion of the investigator
* Patients who have emergent need for starting IV iron
* Patients who will be started on statins within the next 6 weeks
* Patients currently taking PDE5 inhibitors
* Patients allergic to radiocontrast, Zemplar or who can not take nitroglycerin
* Patients known to be HIV positive
* Patients who can not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Richard A. Rodebush VA Medical Center, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Alborzi P, Patel NA, Peterson C, Bills JE, Bekele DM, Bunaye Z, Light RP, Agarwal R. Paricalcitol reduces albuminuria and inflammation in chronic kidney disease: a randomized double-blind pilot trial. Hypertension. 2008 Aug;52(2):249-55. doi: 10.1161/HYPERTENSIONAHA.108.113159. Epub 2008 Jul 7. PMID 18606901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 169 patients screened from renal speciality clinics from November 2006 to June 2007
Period: Overall Study
Arm/Group | 1 | 2 | 3
Started | 8 | 8 | 8
Completed | 7 | 8 | 7
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 | 2 | 3 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 1 | 2 | 5 | 8.0
  >=65 years | 7 | 6 | 3 | 16.0
Age Continuous [Mean (Standard Deviation); unit: years] | 72.6 (9.1) | 67.5 (9.1) | 68.4 (12.4) | 68.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4.0
  Male | 6 | 6 | 8 | 20.0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24.0

OUTCOME MEASURES:

1. Primary Outcome: Anti-Inflammatory Effects of Paricalcitol
Description: change in hsCRP level from baseline to 4 weeks
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: micrograms
Arm/Group | 1 | 2 | 3
Number analyzed (Participants) | 7 | 8 | 7
micrograms | .8 [.3 to 1.9] | .5 [.3 to .9] | 1.5 [1.1 to 2.1]

2. Primary Outcome: Endothelial Protectant Effects of Paricalcitol
Time Frame: 6 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Effect of Paricalcitol on Hypertension
Time Frame: 6 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Effect of Paricalcitol on Kidney Function
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No